CLINICAL TRIAL: NCT03971175
Title: A Prospective, Randomized, Single Blinded Multicentre Trial to Evaluate Molecular Genetic Characterisation of Primary Diagnosed or Relapsed Non Small Cell Lung Cancer by Single or Combination of Diagnostic Procedures
Brief Title: Influence of Biopsy Technique on Moleculargenetic Tumor Characterisation in NSCLC
Acronym: PROFILER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PROFILER study
Record Dates: First submitted 2019-03-11; First posted 2019-06-03 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Pathology, Molecular
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forceps group (Active Comparator)
  Interventions: Procedure: Forceps biopsy
- Cryobiopsy group (Experimental)
  Interventions: Procedure: Cryobiopsy

INTERVENTIONS:
Procedure: Forceps biopsy — Endobronchial biopsy with the forceps
  Arms: Forceps group
Procedure: Cryobiopsy — Endobronchial biopsy with the cryobiopsy probe
  Arms: Cryobiopsy group

SUMMARY:
Study design Prospective multicentre explorative randomized single blinded study to evaluate accuracy of molecular genetic characterisation of NSCLC. Patients with suspected lung cancer are randomized in a 1:1-setting for bronchoscopic tumor tissue either by forceps or by cryobiopsy. Apart from the bronchoscopic techniques liquid biopsy of peripheral blood and if feasible transbronchial needle aspiration with or without endobronchial ultrasound guidance are performed for in all patients.

Objectives

Primary Objective:

assessment of differences in detection of molecular genetic alterations in NSCLC between bronchoscopic forceps biopsy and bronchoscopic cryobiopsy

Secondary Objective:

assessment of differences in detection of molecular genetic alterations in NSCLC between

* liquid biopsy, solid tumor tissue by bronchoscopic techniques, cytologic material by TBNA
* combination of methods (tissue biopsy, TBNA and liquid biopsy) and single techniques
* naïve and processed tumor tissue specimen (eg. microdissection)

To assess differences in side effects e.g. periinterventional bleeding

Explorative Objective:

To explore tumor mutational burden with regard to

* solid tumor tissue by bronchoscopic forceps biopsy by bronchoscopic cryobiopsy
* cytologic material by (EBUS-guided) TBNA
* liquid biopsy

Target subject population Patients with suspected lung cancer or proven NSCLC and visible tumor suspicious lesion(s) requiring tissue diagnosis form the study population of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent to the study and the study specific procedures prior to any study intervention
2. Male or female patients aged ≥18 years
3. Patients with primary diagnosis of suspected lung cancer OR Patients with known NSCLC and suspected relapse after therapy
4. Bronchoscopically visible tumor

Exclusion Criteria:

1. Preexisting malignancy other than NSCLC
2. Contraindication for bronchoscopy according to the international guidelines, daily clinical practice and the local regulations with

   * Patients with existing or at risk of pulmonary and cardiovascular decompensation
   * Patients at increased risk of bleeding with antiplatelet agents except of aspirin (clopidogrel, ticlopidine, …) , anticoagulant therapy (prolonged PTT), thrombocytopenia (< 50.000/ul) or coagulopathy (prolonged in vitro bleeding time).
   * Intolerance to sedation
   * Unstable or immobile cervical spine
   * Limited motion of the temporomandibular joint
3. Previous enrolment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection of at least one molecular and/ or genetic alteration. | recruiting period approximately 24 months
  assessment of differences in detection of molecular genetic alterations in NSCLC between bronchoscopic forceps biopsy and bronchoscopic cryobiopsy
Differences in the detection of total mutational burden between both techniques. | recruiting period approximately 24 months
  assessment of differences in detection of molecular genetic alterations in NSCLC between bronchoscopic forceps biopsy and bronchoscopic cryobiopsy

SECONDARY OUTCOMES:
Detection of any molecular and/ or genetic alterations | recruiting period approximately 24 months
  assessment of differences in detection rate of molecular genetic alterations in NSCLC between
  * different bronchoscopic (forceps/ cryobiopsy) specimens (No 1 to No 4)
  * liquid biopsy, solid tumor tissue by bronchoscopic techniques, cytologic material by TBNA
  * combination of methods (tissue biopsy, TBNA and liquid biopsy) and single techniques
  * naïve and processed tumor tissue specimen (eg. microdissection) To assess differences in side effects e.g. periinterventional bleeding
Combinations of molecular and/ or genetic alterations | recruiting period approximately 24 months
  assessment of differences in detection rate of molecular genetic alterations in NSCLC between
  * different bronchoscopic (forceps/ cryobiopsy) specimens (No 1 to No 4)
  * liquid biopsy, solid tumor tissue by bronchoscopic techniques, cytologic material by TBNA
  * combination of methods (tissue biopsy, TBNA and liquid biopsy) and single techniques
  * naïve and processed tumor tissue specimen (eg. microdissection) To assess differences in side effects e.g. periinterventional bleeding
Differences in the quantity of total mutational burden between the different techniques | recruiting period approximately 24 months
  assessment of differences in the quantity of total mutational burden between
  * different bronchoscopic (forceps/ cryobiopsy) specimens (No 1 to No 4)
  * liquid biopsy, solid tumor tissue by bronchoscopic techniques, cytologic material by TBNA
  * combination of methods (tissue biopsy, TBNA and liquid biopsy) and single techniques
  * naïve and processed tumor tissue specimen (eg. microdissection) To assess differences in side effects e.g. periinterventional bleeding

OTHER OUTCOMES:
Qualitative tumor DNA determination using next generation sequencing techniques for the different specimens | recruiting period approximately 24 months
  to explore tumor mutational burden with regard to
  * Solid tumor tissue by bronchoscopic forceps biopsy by bronchoscopic cryobiopsy
  * Cytologic material by (EBUS-guided) TBNA
  * Liquid biopsy
Quantitative tumor DNA determination using next generation sequencing techniques for the different specimens | recruiting period approximately 24 months
  to explore tumor mutational burden with regard to
  * Solid tumor tissue by bronchoscopic forceps biopsy by bronchoscopic cryobiopsy
  * Cytologic material by (EBUS-guided) TBNA
  * Liquid biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Tübingen, Germany